CLINICAL TRIAL: NCT03005886
Title: The Effect of Periodontal Therapy on Neopterin and Vascular Cell Adhesion Molecule-1 Levels in Chronic Periodontitis Patients With and Without Acute Myocardial Infarction
Brief Title: The Effect of Periodontal Therapy in Chronic Periodontitis Patients With and Without Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Research Assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 03/2006-30
Record Dates: First submitted 2016-12-20; First posted 2016-12-30 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Myocardial Infarction; Chronic Periodontitis
Keywords: Periodontitis; Periodontal-systemic disease; Cardiovascular diseases; Gingival crevicular fluid; Acute myocardial infarction; Neopterin; Vascular cell adhesion molecule-1
MeSH Terms: conditions — Myocardial Infarction; Chronic Periodontitis; Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AMI+CP: (Experimental): GCF sampling,periodontal examination,phase I therapy:
  Patients, who met the AMI diagnostic criteria with chronic periodontitis. Baseline periodontal examination of AMI patients and 24-48h GCF sampling was carried out in their hospital bed under sufficient illumination using artificial light. Phase I periodontal therapy including comprehensive proper plaque control program, scaling, subgingival curettage and root planning in Department of Periodontology. Mucoperiosteal flap operation was performed in cases where needed.
  Interventions: Procedure: Periodontal examination; Procedure: GCF sampling; Procedure: phase I therapy
- Chronic Periodontitis (CP) (Active Comparator): GCF sampling,periodontal examination,phase I therapy:
  Systemically healthy chronic periodontitis patients.Phase I periodontal therapy including comprehensive proper plaque control program, scaling, subgingival curettage and root planning in Department of Periodontology.Mucoperiosteal flap operation was performed in cases where needed.
  Interventions: Procedure: Periodontal examination; Procedure: GCF sampling; Procedure: phase I therapy
- Healthy controls (Sham Comparator): clinically healthy individuals not having any periodontal and systemic diseases history.Comprehensive medical and periodontal examination to confirm that they did not have systemic and periodontal diseases
  Interventions: Procedure: Periodontal examination; Procedure: GCF sampling

INTERVENTIONS:
Procedure: Periodontal examination — periodontal examination included the assessment of plaque index (PI), gingival index(GI), probing depth (PD), bleeding on probing (BOP) and clinical attachment level (CAL).
  All subjects underwent a periodontal examination performed by the same periodontitis (ZTÇ) Prior to the study, the examiner was calibrated for reproducibility of PD and CAL measurements
Procedure: GCF sampling — GCF samples were collected using commercially available periopaper . The sample site was gently air-dried and all supragingival plaque was removed. The area was carefully isolated with cotton rolls and a saliva ejector was used to prevent the samples from being contaminated by saliva. The paper strips were inserted into the pockets until slight resistance was felt and left in place for 30s.
Procedure: phase I therapy — comprehensive proper plaque control program, scaling, subgingival curettage and root Phase I Periodontal Therapy planning
  Arms: AMI+CP:; Chronic Periodontitis (CP)

SUMMARY:
The aim of this study was to evaluate the effects of periodontal treatment on gingival crevicular fluid (GCF) levels of Neopterin(N) and vascular cell adhesion molecule (VCAM-1) in chronic periodontitis(CP) patients with acute myocardial infarction(AMI) in comparison to systemically healthy CP patients. The investigators' hypothesized that severe CP may play a role in initiating or exacerbating MI and there is an increased risk for AMI among systemically healthy persons affected with severe CP.

DETAILED DESCRIPTION:
There are no studies specifically addressing the altered GCF profile concurrent with the onset of myocardial infarction acutely (i.e. in the first 24h) and no data are currently available about GCF Neopterin and VCAM-1 levels in AMI patients with chronic periodontitis. The present study aimed to assess whether GCF levels of CP patients with AMI have an alteration in GCF levels of Neopterin and VCAM-1, also assessed whether these alterations might be related to treatment of existing periodontitis in AMI patients. A total of 60 subjects (20 CP patients with AMI, 20 systemically healthy CP patients and 20 healthy controls) were included.GCF samples were analyzed baseline and after 3 and 6 months, probing pocket depth(PD), clinical attachment level (CAL),bleeding on probing (BOP) , gingival and plaque (PI) indices were recorded. Neopterin and VCAM-1 levels (concentration and total amount) were determined by enzyme linked immunosorbent assay (ELISA). Baseline periodontal examination of AMI patients and 24-48h GCF collection was carried out in their hospital bed under sufficient illumination using artificial light. Within a time period of 2 months after the proceeding infarction, none of the patients had received periodontal treatment. AMI patients underwent periodontal therapy after the stabilization of their condition with the consent from same cardiologist. Periodontal disease was diagnosed based on the 1999 classification system developed by Armitage, and a preoperative periapical radiograph was taken that provided baseline data in Faculty of Dentistry. Clinical index scores and GCF sampling were recorded before, 3 and 6 months after the periodontal treatment. All selected patients underwent a 2- to 4-week initial therapy, which included comprehensive proper plaque control program, scaling, subgingival curettage and root planning in Department of Periodontology. In all patients a periodontal reevaluation was performed 4 weeks after phase I therapy, to confirm the suitability of the sites for periodontal surgery. Mucoperiosteal flap operation was performed in cases where needed. The blood samples for serum were centrifuged for 10 min at 11.00RPM separating the serum from the cells. The serum samples were then immediately divided into 0.2-0.5ml aliquots and stored at -80°C until required for analysis. Samples were assayed for N and VCAM-1 using quantitative enzyme immunoassays.

Micro-centrifuge tubes, containing periopaper strips with absorbed GCF sample, were allowed to reach room temperature and eluted using a centrifugal method.17 After centrifugation, the strips were removed and the fluid was assayed by ELISA for N and soluble VCAM-1.The levels of N and sVCAM-1 in serum and GCF samples were measured using ELISA kit , . The ELISA procedures were carried out according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* None of the patients had received periodontal treatment during the past 6 months and none had received antibiotic medication during the past 3 months.
* AMI+CP and CP groups were regarded as suitable for the study if they were affected by CP and had at least 16 teeth, including at least four molars in different quadrants at least two periodontal pocket at least 5mm in depth, with a minimum of 2mm attachment loss.
* Patients, who met the AMI diagnostic criteria, with or without persistent ST-segment elevation

Exclusion Criteria:

* Patients with neoplasias, liver cirrhosis, HIV infection, chronic renal failure, hypo or hyperparathyroidism, diabetes mellitus, chronic inflammatory diseases (rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, and Chron's Disease

Ages: 39 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Concentration and total amount of serum and GCF VCAM-1 and Neopterin | Change from baseline concentration and total amount of serum&GCF sVCAM-1 and Neopterin at 6months.
  Using the standards included with the Enzyme-Linked ImmunoSorbent Assay (ELISA) kit. The concentrations of Neopterin and sVCAM-1 were expressed as ng/ml. Total amounts were also calculated by multiplying concentrations and GCF volumes(ml) and expressed as ng.

SECONDARY OUTCOMES:
Clinical attachment level(CAL) | Baseline, 3 and 6 months after initial periodontal treatment
  CAL was calculated as the distance from cemento-enamel junction to bottom of gingival sulcus.

OTHER OUTCOMES:
Plaque Index | Baseline, 3 and 6 months after initial periodontal treatment
  Plaque Index were calculated as a sum of mean scores by each examined tooth divided by the number of evaluated teeth.
Gingival Index | Baseline, 3 and 6 months after initial periodontal treatment
  Gingival Index were calculated as a sum of mean scores by each examined tooth divided by the number of evaluated teeth.
Probing Depth | Baseline, 3 and 6 months after initial periodontal treatment
  PD was recorded as the distance from the gingival margin to the most apical part of the sulcus.
Bleeding on probing | Baseline, 3 and 6 months after initial periodontal treatment
  BOP is a widely used criterion to diagnose inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Turgut Çankaya, PhD DDs, Principal Investigator — Gazi University; Ayşen Bodur, PhD DDS, Study Director — Gazi University

IPD SHARING:
Plan to Share IPD: Yes
Clinical measurement records of periodontal and medical protocols can be shared with other researches. Researches should send an e-mail to principal investigator.
Supporting Information: SAP
Time Frame: The data will become available after the study paper published for one year period.
Access Criteria: The statistical analysis in the published paper will be shared